CLINICAL TRIAL: NCT05984043
Title: Piloting a Biofeedback Intervention for Adolescents With Overweight and a History of Adverse Childhood Experiences
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution without completing this trial. No participants enrolled.
Sponsor: Colorado State University (Other)
Collaborators: Children's Hospital Colorado (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5P30DK048520-29 (NIH)
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity | interventions — Biofeedback, Psychology; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Waitlist (Other)
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: Biofeedback — Heart-rate Variability Biofeedback
  Arms: Biofeedback
Other: Waitlist — Waitlist control group
  Arms: Waitlist

SUMMARY:
Adverse childhood experiences (ACEs), referring to traumatic experiences occurring before 18 years of age (e.g., abuse/neglect), are associated with a 30-70% increased risk of developing adolescent and adult obesity and obesity-related cardiometabolic comorbidities, which may be due to dysregulation in stress-related physiology and engagement in stress-related behaviors. While adolescents with ACEs have a 2.25 times increased risk of obesity, standard-of-care lifestyle (e.g., nutrition/physical activity) interventions do not typically incorporate trauma-informed care, including assessment and therapeutic attention to effects of ACEs. Heart rate variability (HRV) biofeedback is an evidence-based, relatively brief, mind-body intervention targeting the stress physiology that can be dysregulated in adolescents with ACEs. The objective of this proposal is to adapt and test a 4-session HRV biofeedback protocol for 12-17-year-olds with BMI>85th percentile and ACEs. First (Phase 1), we will iteratively adapt a 4-session HRV biofeedback facilitator protocol with n=3-5 adolescents with overweight/obesity and ACEs, using adolescent quantitative and qualitative feedback to hone and optimize HRV biofeedback for this population (Aim 1). Next (Phase 2), we will conduct a randomized waitlist-controlled pilot study of n=30 adolescents with overweight/obesity and ACEs to assess acceptability and feasibility (Aim 2) and to describe changes in theorized targets of biofeedback (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Four or more ACEs
* BMI at or above the 85th percentile;

Exclusion Criteria:

* Major renal, hepatic, endocrinologic, rheumatologic, cardiac, or pulmonary medical problem likely to affect mood or weight
* Medications affecting mood or weight (e.g. anti-anxiety/depressants/psychotics, stimulants, mood stabilizers, insulin sensitizers, weight loss)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Facilitator Protocol | Year 1
  4-session biofeedback facilitator protocol
Feasibility/Acceptability | Year 1
  Protocol implementation will be feasible in terms of recruitment (≥60% eligible enroll), intervention adherence (≥80% will receive >80% dosage), baseline/post-treatment assessment adherence (<20% missing data), and post-treatment retention (≥80%). Biofeedback will be acceptable based on session likeability ratings (80% >4:5) and qualitative themes assessed by interview indicative of likeability/benefit.
Stress Physiology | Year 2
Stress Eating | Year 2
Inflammatory Biomarkers | Year 2
Insulin Sensitivity | Year 2

IPD SHARING:
Plan to Share IPD: No